CLINICAL TRIAL: NCT06035692
Title: Effect of Brachial Plexus Block on Outcomes of Upper Extremity Arteries After Intracranial Aneurysm Interventional Surgery Via Transradial Access: A Randomized Clinical Trial
Brief Title: Application of Brachial Plexus Block in Patients Undergoing Cerebral Aneurysm Embolization Via Transradial Approach
Acronym: ABPBCAETRA
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The First Affiliated Hospital with Nanjing Medical University (Other)
Collaborators: Xuzhou Central Hospital (Other); Huizhou Municipal Central Hospital (Other); Nanjing Jiangbei Hospital (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: BPB
Record Dates: First submitted 2023-06-27; First posted 2023-09-13 (Actual); Last update posted 2024-02-28 (Actual); Status verified 2024-02

CONDITIONS: Intracranial Aneurysm; Transradial Access(TRA)
MeSH Terms: conditions — Intracranial Aneurysm | interventions — Ropivacaine; Brachial Plexus Block

STUDY DESIGN:
Intervention Model Description: This is a multicenter prospective randomized controlled study.Patients were assigned to the two groups with the use of central randomization and competitive enrollment.
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: In this study, participants, data recorders(investigators), and outcome assessor were unaware of group assignments.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Brachial plexus block group（BPB） (Experimental): All patients received receive Ultrasound-guided BPB with 0.15% ropivacaine 20ml 30min before surgery
  Interventions: Drug: Ropivacaine
- Control group （Control） (No Intervention): All patients received receive Ultrasound-guided BPB with normal saline 20ml 30min before surgery

INTERVENTIONS:
Drug: Ropivacaine — According to the results of the preliminary experiment, the BPB group was given ultrasound-guided BPB with 0.15% ropivacaine 20ml.The ropivacaine concentration was the 90% minimum effective concentration(MEC90) for preventing vasospasm during operation.
  Other Names: brachial plexus block
  Arms: Brachial plexus block group（BPB）

SUMMARY:
The aim of this study was toinvestigate the effect of BPB on outcome of upper extremity arteries in patients undergoing interventional embolization of intracranial aneurysms via TRA. A multicenter prospective clinical trial was designed. The study subjects were patients undergoing cerebral aneurysm embolization with TRA. BPB was given in the BPB group patients and no BPB in the control group.The incidence of radial artery spasm (RAS) diagnosed by intraoperative angiography and the occurrence of the unfavorable RA for repeated trans-radial interventions (TRI) diagnosed by vascular ultrasound 1 month after surgery， perioperative changes of blood flow parameters in upper limb vessels,postoperative inflammatory factors and complications were observed in the two groups.

DETAILED DESCRIPTION:
The aim of this study was to investigate the effect of BPB on outcome of upper extremity arteries in patients undergoing interventional embolization of intracranial aneurysms via TRA. A multicenter prospective clinical trial was designed, and the study subjects were patients undergoing cerebral aneurysm embolization with TRA. Participants were randomly assigned to receive Ultrasound-guided BPB with 0.15% ropivacaine 20ml (BPB group) or normal saline 20ml (Control group) in 1:1ratio.The primary outcomes measured were the incidence of RAS diagnosed by intraoperative angiography and the occurrence of the unfavorable RA for repeated trans-radial interventions (TRI) diagnosed by vascular ultrasound 1 month after surgery.Secondary outcomes included the severity of RAS, Components of unfavorable RA for repeated TRI, intraoperative nitroglycerin use, Intraoperative hypotension, surgeon satisfaction scores.

ELIGIBILITY:
Inclusion Criteria:

* 18-75 years old, BMI<28kg/m2
* ASA physical status Ⅰ-Ⅲ
* Elective interventional surgery for intracranial aneurysms via TRA
* willing to sign informed consent

Exclusion Criteria:

* patients allergic to local anesthetics
* neck infection on the surgical side
* Preoperative upper extremity ultrasound or DSA showed radial artery occlusion and arteriovenous fistula
* The diameter of radial artery was still less than 2mm after brachial plexus block
* Axillary artery occlusion and other vascular anatomical abnormalities may affect the operation
* Radial artery patency: Barbeau type D
* The history of hand trauma may affect the establishment of radial artery; access, or the use of radial artery as a bypass or dialysis vessel
* patients with incomplete block effect after nerve block were detected;
* The patient refused to participate in the study or cooperate with the follow-up

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 176 (Estimated)
Dates: Start 2023-06-01 (Actual); Primary Completion 2024-02-29 (Estimated); Study Completion 2024-06-30 (Estimated)

PRIMARY OUTCOMES:
Assess the RAS by angiography at the begining of the operation | During the operation
  The RAS was assessed through radial artery angiography following the insertion of the arterial catheter.
Evaluate the degree of RAS by angiography at the end of the operation | During the operation
  The severity of RAS was classified as severe, moderate, or mild based on the degree of stenosis observed on radial arteriography: greater than 75%, 25-75%, and less than 25% of the vessel diameter, respectively. In addition, if the combined spasm length exceeded 2cm, the severity increased by 1 grade.

SECONDARY OUTCOMES:
Assess unfavorable RA for repeated trans-radial interventions (TRI) at 1 month after surgery by ultrasonography. | Month 1 after surgery
  The the radial artery was evaluated at 1 month after surgery using ultrasonography by an anesthesiologist who was blinded to the group assignments.The radial artery was considered unfavorable for repeated-TRI if it exhibited any of the following criteria: total occlusion, intima-media thickness (IMT) ≥0.5 mm and diameter <1.5mm, moderate and diffuse stenosis (> 10 mm in length), or severe focal or diffuse stenosis (regardless of length).
Record the incidence of intima-media thickness (IMT) ≥0.5 mm and diameter <1.5mm at 1 month after surgery by ultrasonography. | Month 1 after surgery
  The incidence of intima-media thickness (IMT) ≥0.5 mm and diameter <1.5mm as a component of unfavorable RA for repeated TRI was recorded at one month follow-up.
Record the incidence of radial artery occlusion at 1 month after surgery by ultrasonography. | Month 1 after surgery
  The incidence of radial artery occlusion as a component of unfavorable RA for repeated TRI was recorded at one month follow-up.
Record the incidence of moderate and diffuse stenosis (> 10 mm in length) at 1 month after surgery by ultrasonography. | Month 1 after surgery
  The incidence of moderate and diffuse stenosis (> 10 mm in length) as a component of unfavorable RA for repeated TRI was recorded at one month follow-up.
Record the incidence of severe focal or diffuse stenosis (regardless of length) at 1 month after surgery by ultrasonography. | Month 1 after surgery
  The incidence of severe focal or diffuse stenosis (regardless of length) as a component of unfavorable RA for repeated TRI was recorded at one month follow-up.
Record the use of nitroglycerin during the operation | During the operation
  When the radial sheath was inserted, upper limb angiography was performed, and nitroglycerin 200ug was administered if any degree of vasospasm in the upper limb was observed on the angiography. The administration of nitroglycerin in each group was recorded.
Record the incidence of intraoperative hypotension | During the operation
  The definition of intraoperative hypotension was a mean arterial blood pressure below 60mmHg.
Record physician satisfaction by questionnaire | Day 0 after the surgery
  Physician satisfaction was scored on a scale of 1-10, with a score of 1 indicating very poor and dissatisfied experience and a score of 10 indicating very satisfied. The surgeons were asked to fill in the satisfaction questionnaire according to the operation situation after operation and recorded.
Record the duration of radial artery puncture | At the begining of the operation
  The time from the beginning of the radial artery puncture to the placement of the radial sheath was recorded.
Measured diameter and the hemodynamic parameters of radial artery by ultrasound 30min after BPB or control interventions | 30min after BPB or control interventions
  The radial artery was evaluated(include diameter, PSV,EDV,TAMAX,PI,RI) before the surgery using ultrasonography by an anesthesiologist who was blinded to the group assignments.
Measured diameter and the hemodynamic parameters of radial artery by ultrasound 24h after surgery | 24h after surgery
  The radial artery was evaluated(include diameter, PSV,EDV,TAMAX,PI,RI) before the surgery using ultrasonography by an anesthesiologist who was blinded to the group assignments.
Measured diameter and the hemodynamic parameters of radial artery by ultrasound 1 month after surgery | Month 1 after surgery
  The radial artery was evaluated(include diameter, PSV,EDV,TAMAX,PI,RI) before the surgery using ultrasonography by an anesthesiologist who was blinded to the group assignments.
Measured diameter and the hemodynamic parameters of ulnar artery by ultrasound 30min after BPB or control interventions | 30min after BPB or control interventions
  The ulnar artery was evaluated(include diameter, PSV,EDV,TAMAX,PI,RI) before the surgery using ultrasonography by an anesthesiologist who was blinded to the group assignments.
Measured diameter and the hemodynamic parameters of ulnar artery by ultrasound 24h after surgery | 24h after surgery
  The ulnar artery was evaluated(include diameter, PSV,EDV,TAMAX,PI,RI) before the surgery using ultrasonography by an anesthesiologist who was blinded to the group assignments.
Measured diameter and the hemodynamic parameters of ulnar artery by ultrasound 1 month after surgery | Month 1 after surgery
  The ulnar artery was evaluated(include diameter, PSV,EDV,TAMAX,PI,RI) before the surgery using ultrasonography by an anesthesiologist who was blinded to the group assignments.
Measured diameter and the hemodynamic parameters of brachial artery by ultrasound 30min after BPB or control interventions | 30min after BPB or control interventions
  The brachial artery was evaluated(include diameter, PSV,EDV,TAMAX,PI,RI) before the surgery using ultrasonography by an anesthesiologist who was blinded to the group assignments.
Measured diameter and the hemodynamic parameters of brachial artery by ultrasound 24h after surgery | 24h after surgery
  The brachial artery was evaluated(include diameter, PSV,EDV,TAMAX,PI,RI) before the surgery using ultrasonography by an anesthesiologist who was blinded to the group assignments.
Measured diameter and the hemodynamic parameters of brachial artery by ultrasound 1 month after surgery | Month 1 after surgery
  The brachial artery was evaluated(include diameter, PSV,EDV,TAMAX,PI,RI) before the surgery using ultrasonography by an anesthesiologist who was blinded to the group assignments.
Record mean arterial pressure at different time points | During the operation
  The mean intraoperative arterial pressure from T0 to T8 was recorded. T0 indicates time after entering the operating room; T1,30 minutes after BPB or control procedure; T2, 5 minutes after induction of general anesthesia; T3, angiography after the radial sheath enters the radial artery; T4,1minutes after angiography; T5, 3minutes after angiography; T6, 5minutes after angiography; T7, 10 minutes after angiography; T8, completion of the operation.
Record perioperative complications | Day 1 after the surgery
  Perioperative complications include puncture site complications, brachial plexus complications, and other cardiovascular and cerebrovascular complications
Recorded the levels of eight inflammatory factors | Day 1 after the surgery
  The hospital laboratory conducted an examination on 8 inflammatory factors (include IL-2,IL-4,IL-6,IL-10,IL-17,IL-12P70,IFN-r,TNF-a) to assess postoperative infection, and subsequently provided the results.
Recorded the incidence of postoperative acute embolism events | Day 1 after the surgery
  A head magnetic resonance imaging(MRI) was conducted to document the occurrence of postoperative embolic events, such as acute cerebral infarction.

OTHER OUTCOMES:
Calculate MEC50 and MEC95 of ropivacaine in brachial plexus block by sequential method | During the operation
  The minimum effective concentration（MEC50 and MEC90） of ropivacaine for brachial plexus block to prevent radial artery spasm during operation was determined by sequential method.
Record diameter and the hemodynamic parameters of radial artery by ultrasound | Day 1 before surgery
  The radial artery was evaluated(include diameter, PSV,EDV,TAMAX,PI,RI) before the surgery using ultrasonography by an anesthesiologist who was blinded to the group assignments.
Record diameter and the hemodynamic parameters of brachial artery by ultrasound | Day 1 before surgery
  The brachial artery was evaluated(include diameter, PSV,EDV,TAMAX,PI,RI) before the surgery using ultrasonography by an anesthesiologist who was blinded to the group assignments.
Record diameter and the hemodynamic parameters of ulnar artery by ultrasound | Day 1 before surgery
  The ulnar artery was evaluated(include diameter, PSV,EDV,TAMAX,PI,RI) before the surgery using ultrasonography by an anesthesiologist who was blinded to the group assignments.

CONTACTS AND LOCATIONS:
Overall Officials: Jingjin Li, M.D, Principal Investigator — The First Affiliated Hospital with Nanjing Medical University
Locations (1):
- The First Affiliated Hospital with Nanjing Medical University, Nanjing, Jiangsu, China

IPD SHARING:
Plan to Share IPD: Yes
If anyone is interested in this study, please contact us, and I think we would like to share IPD with him
Supporting Information: Study Protocol, CSR
Time Frame: Month 1
Access Criteria: If anyone is interested in this study, please contact us, and I think we would like to share IPD with him